CLINICAL TRIAL: NCT07231952
Title: A Phase II Study of Time-limited Combination of Pirtobrutinib, Venetoclax, and Rituximab in Treatment Naïve Patients With Waldenström's Macroglobulinemia (WM) / Lymphoplasmacytic Lymphoma (LPL) (PRoVen)
Brief Title: A Study of Pirtobrutinib, Venetoclax, and Rituximab in People With Waldenström's Macroglobulinemia (WM)/Lymphoplasmacytic Lymphoma (LPL)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: AbbVie (Industry); Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 25-149
Record Dates: First submitted 2025-11-13; First posted 2025-11-17 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Waldenstrom Macroglobulinemia; Lymphoplasmacytic Lymphoma
Keywords: Waldenstrom Macroglobulinemia; Lymphoplasmacytic Lymphoma; Memorial Sloan Kettering Cancer Center; 25-149
MeSH Terms: conditions — Waldenstrom Macroglobulinemia; Lymphoma, B-Cell, Marginal Zone | interventions — pirtobrutinib; venetoclax; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Participants with Waldenström's Macroglobulinemia (WM)/Lymphoplasmacytic Lymphoma (LPL) (Experimental): Participants with treatment naive Waldenström's Macroglobulinemia (WM)/Lymphoplasmacytic Lymphoma (LPL)
  Interventions: Drug: Pirtobrutinib; Drug: Venetoclax; Drug: Rituximab

INTERVENTIONS:
Drug: Pirtobrutinib — PO QD
Drug: Venetoclax — PO QD
Drug: Rituximab — IV or SC

SUMMARY:
The purpose of this study is to find out if the combination of pirtobrutinib, venetoclax, and rituximab is an effective treatment for participants with Waldenström's macroglobulinemia (WM)/lymphoplasmacytic lymphoma (LPL)

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18 years
* Histologically confirmed treatment naive WM/LPL
* Patients must have measurable disease as defined by at least one lymph node ≥1.5 cm and/ or IgM levels > 0.5gm/dl quantified by using densitometry on serum protein electrophoresis (SPEP) or quantitative nephelometry.
* Participants must have at least one of the established criteria to require therapy for WM, including anemia, thrombocytopenia, neuropathy related to WM, symptomatic hyperviscosity or serum viscosity levels greater than 4.0 centipoises, WM-associated glomerulonephritis or renal disease, bulky disease, or constitutional symptoms
* ECOG performance status ≤2
* Platelet count ≥ 50,000 cells/mm3, independent of transfusions within 7 days of screening assessment
* Hemoglobin ≥ 8 g/dL, unless due to disease involvement in which case ≥ 7 g/dL, independent of transfusions within 7 days of screening assessment
* Absolute neutrophil count >1000 cells/mcL, independent of growth factor support within 7 days of screening assessment
* Total bilirubin < 1.5 x upper normal institutional limits. In patients with Gilbert's disease total bilirubin up to 3x ULN will be allowed
* AST(SGOT)/ALT(SGPT) < 3 x institutional upper limit of normal unless elevation is caused by liver involvement with WM in which case AST and ALT may be ≤ 5 x ULN
* Creatinine within normal institutional limits OR Creatinine clearance >40 mL/min for patients with creatinine levels above institutional normal (by Cockcroft-Gault estimate or 12-24h creatinine clearance measurements)
* Adequate coagulation, defined as activated partial thromboplastin time (aPTT) or partial thromboplastin time (PTT) and prothrombin (PT) or (international normalized ratio (INR) not greater than 1.5 x ULN
* Ability to understand and the willingness to sign a written informed consent document.
* Patient must be able to swallow pills
* Patients with Hepatitis B surface antibody serum positivity due to prior immunization, as well as those with Hepatitis B core antibody positivity with negative PCR on antiviral therapy will be eligible.
* Willingness of participants of reproductive potential and their partners to observe highly effective birth control methods for the duration of treatment and for 1 year following the last dose of study treatment

Exclusion Criteria:

* Prior/Concomitant Therapy: Participants must not have had prior systemic therapy.
* Medical Conditions

  * Major surgery within 4 weeks prior to start of treatment
  * History of bleeding diathesis
  * Patients who experienced a major bleeding event or grade ≥ 3 arrhythmia on prior treatment with a BTK inhibitor.
  * NOTE: Major bleeding is defined as bleeding having one or more of the following features: potentially life-threatening bleeding with signs or symptoms of hemodynamic compromise; bleeding associated with a decrease in the hemoglobin level of at least 2g per deciliter; or bleeding in a critical area or organ (e.g., retroperitoneal, intraarticular, pericardial, epidural, or intracranial bleeding or intramuscular bleeding with compartment syndrome)
  * History of stroke or intracranial hemorrhage within 6 months of start of treatment
  * History of allogeneic or autologous stem cell transplant (SCT) or chimeric antigen receptor-modified T-cell (CAR-T) therapy within 60 days of start of treatment or presence of any of the following, regardless of prior SCT and/or CAR-T therapy timing:
  * active graft versus host disease (GVHD);
  * cytopenia from incomplete blood cell count recovery post-transplant;
  * need for anti-cytokine therapy for toxicity from CAR-T therapy; residual symptoms of neurotoxicity > Grade 1 from CAR-T therapy;
  * ongoing immunosuppressive therapy (> 20 mg prednisone or equivalent daily).
* Significant cardiovascular disease defined as:

  * unstable angina or acute coronary syndrome within the past 2 months prior to start of treatment
  * history of myocardial infarction within 3 months prior to start of treatment or
  * documented LVEF by any method of ≤ 40% in the 12 months prior to start of treatment
  * ≥ Grade 3 NYHA functional classification system of heart failure
  * Uncontrolled or symptomatic arrhythmias
* Prolongation of the QT interval corrected for heart rate (QTcF) > 470 msec. QTcF is calculated using Fridericia's Formula (QTcF): QTcF = QT/(RR0.33).

  * Correction of suspected drug-induced QTcF prolongation can be attempted at the investigator's discretion and only if clinically safe to do so with either discontinuation of the offending drug or switch to another drug not known to be associated with QTcF prolongation.
  * Correction for underlying bundle branch block (BBB) allowed. Note: Patients with pacemakers are eligible if they have no history of fainting or clinically relevant arrhythmias while using the pacemaker
* Patients who have tested positive for Human Immunodeficiency Virus (HIV) are excluded due to risk of opportunistic infections with both HIV and BTK- inhibitors. For patients with unknown HIV status, HIV testing will be performed at Screening and result must be negative for enrollment.
* Known active hepatitis B virus (HBV) or hepatitis C virus (HCV) infection based on criteria below:

  * Hepatitis B virus (HBV):
  * Patients with positive hepatitis B surface antigen (HBsAg) are excluded.
  * Patients with positive hepatitis B core antibody (anti-HBc) and negative HBsAg require a negative hepatitis B polymerase chain reaction (PCR) evaluation before start of treatment.
  * Patients who are HBV DNA PCR positive will be excluded.
  * Hepatitis C virus (HCV): positive hepatitis C antibody. If positive hepatitis C antibody result, patient will need to have a negative result for hepatitis C ribonucleic acid (RNA) before start of treatment. Patients who are hepatitis C RNA positive will be excluded.
* Known active cytomegalovirus (CMV) infection. Unknown or negative status are eligible.
* Pregnancy or plan to become pregnant during the study or within 1 month of the last dose of study treatment.
* Lactation or plan to breastfeed during the study or within 1 week of the last dose of study treatment.
* Clinically significant active malabsorption syndrome or other condition likely to affect gastrointestinal (GI) absorption of the study drug.
* Evidence of other clinically significant uncontrolled condition(s) including but not limited to, uncontrolled systemic bacterial, viral, fungal or parasitic infection (except for fungal nail infection), or other clinically significant active disease process which in the opinion of the investigator and medical monitor may pose a risk for patient participation. Screening for chronic conditions is not required.
* Active uncontrolled auto-immune cytopenia (e.g., autoimmune hemolytic anemia [AIHA], idiopathic thrombocytopenic purpura [ITP]) for which new therapy was introduced or existing therapy was escalated within the 4 weeks prior to study enrollment to maintain adequate blood counts.
* Active second malignancy unless in remission and with life expectancy > 2 years.
* Patients requiring therapeutic anticoagulation with warfarin or another vitamin K antagonist.
* Vaccination with live vaccine within 28 days prior to start of treatment
* Other Exclusions

  * Have a known hypersensitivity to any of the excipients of Pirtobrutinib or to any intended study medications.
  * Participants who require ongoing use or received a moderate or strong CYP3A inducer, moderate or strong CYP3A inhibitor, P-gp inhibitor within 7 days prior to the first dose of study drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-11-11 (Actual); Primary Completion 2028-04-11 (Estimated); Study Completion 2028-04-11 (Estimated)

PRIMARY OUTCOMES:
Number of participants with Very Good Partial Response Rate or Better | 1 year
  To evaluate the rate of very good partial response (VGPR) rate or better in previously untreated participants with WM / LPL who are treated upfront with this regimen.

CONTACTS AND LOCATIONS:
Overall Officials: M. Lia Palomba, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (8):
- United States (8):
  - Beth Israel Deaconess Medical Center (Data Collection Only), Boston, Massachusetts
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Memoral Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Memorial Sloan Kettering Suffolk - Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org